CLINICAL TRIAL: NCT02808130
Title: A CASE CONTROL STUDY TO DETERMINE THE GINGIVAL CREVICULAR FLUID MALONDIALDEHYDE, PROTEIN CARBONYL AND TOTAL ANTIOXIDANT CAPACITY IN PATIENTS WITH PERIODONTAL DISEASE AND HYPERLIPIDEMIA
Brief Title: PERIODONTAL DISEASE AND HYPERLIPIDEMIA
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, muge lutfioglu, ASSOC PROF, Ondokuz Mayıs University
Other Study IDs: OMU KAEK 2012/43-0.06.12
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Hyperlipidemia, Periodontitis, Gingivitis
Keywords: hyperlipidemia, periodontal disease, oxidative stress,
MeSH Terms: conditions — Hyperlipidemias; Periodontitis; Gingivitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid

GROUPS / COHORTS (6):
- group H: Group H: normolipidemic+ periodontally healthy individuals The healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis
- Group G: Group G: normolipidemic + gingivitis individuals the healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis
- Group CP: Group CP: normolipidemic + generalized chronic periodontitis individuals the healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis
- Group HH: Group HH: hyperlipidemic + periodontally healthy individuals Hyperlipidemia was defined as the presence of one or more altered values of the lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis
- Group HG: Group HG: hyperlipidemic + gingivitis individuals Hyperlipidemia was defined as the presence of one or more altered values of the lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis
- group HCP: Group HCP: hyperlipidemic + generalized chronic periodontitis individuals Hyperlipidemia was defined as the presence of one or more altered values of the lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  Interventions: Other: hyperlipidemia, periodontitis, gingivitis

INTERVENTIONS:
Other: hyperlipidemia, periodontitis, gingivitis — GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva

SUMMARY:
The investigators hypothesized that hyperlipidemia as an unfavourable levels of lipoprotein subfractions have deleterious impact on the development of periodontal infection by altering oxidative stres status of periodontal tissues. The aim of this study was therefore to investigate i) effect of hyperlipidemia on oxidative change in GCF content, ie. MDA, PC and TAOC levels in patients with different periodontal status,

DETAILED DESCRIPTION:
An observational study was performed in 45 hyperlipidemic(22 females, 23 males) and 45 age and sex matched normolipidemic (25 females, 20 males) healthy controls. The participants were recruited as a joint collaboration between Periodontology Department of the Faculty of Dentistry and the Endocrinology and Metabolic Diseases Department of the Faculty of Medicine at Ondokuz Mayis University in Samsun, Turkey between january 2013 and august 2014.The study protocol was approved by the Local Ethics Committee, and written informed consent was obtained from all study participants in accordance with the Helsinki Declaration (revised in 2000) It has been asserted that elevated serum lipid levels create a pro-inflammatory state, which leads to an increase in oxidative state by composing an imbalanced production between highly reactive molecular species and antioxidant defences, consequently predisposing one to infections. Hyperlipidemia claimed to lead an increase in production of reactive oxygen species (ROS) and lipid peroxidation (LPO). On the other hand it has been suggested that high-cholesterol diet increases OS and causes oxidative damage in various organs. Also, OS related mediators have frequently shown to be associated with chronic periodontitis (CP) related inflammatory responses . Excessive ROS derived radical formations reported to have an important role in the inflammatory process by leading to damage to proteins, DNA, carbohydrates, and lipids.

Hyperlipidemia was defined as the presence of one or more altered values of the lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl).

Periodontal status was determined by evaluating the following clinical parameters: Silness & Löe plaque index ; Löe & Silness gingival index ; Probing pocket dept,clinical attachment level, bleeding on probing (BOP) measurements were performed on 6 sites per tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual) using a Williams periodontal probe. GCF collection was subsequently performed using those sites that fit the criteria for GCF sampling described below.

All samples were collected between 8-10 am on the day following periodontal status assessment. Samples were collected from the deepest 6 sites in the chronic periodontitis group. In the gingivitis group samples were collected from the teeth with bleeding on probing, whereas teeth without BOP were chosen in the healthy group. GCF samples were collected from the similar 6 sites in the gingivitis and periodontally healthy groups in order to maintain consistency of sampling. Accordingly, total of 90 GCF samples were taken from each of the 6 groups (15 individuals per group x 6 sites).

ELIGIBILITY:
Inclusion Criteria:

(i) ≥ 18 years of age and having ≥ 16 teeth; (ii)no periodontal therapy in the 6 months prior to data collection; (iii) no systemic problems or chemotherapy within the 6 weeks prior to data collection and any anti-lipaemic drug treatment; (iv) no previous history of smoking.

Exclusion Criteria:

(i) medical history of cancer, rheumatoid arthritis, diabetes mellitus, or cardiovascular disease and any other systemic disease affecting lipid metabolism(i.e. impaired glucose tolerance, metabolic syndrome); (ii) compromised immune system; (iii) pregnancy, menopause, or lactation; (iv) ongoing drug therapy that might affect the clinical characteristics of periodontitis and lipid metabolism; (v) use of systemic antimicrobials during the 6 weeks prior to data collection; and (vi) dental treatment during the 6 months prior to data collection.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: An observational case-control study was performed in 45 hyperlipidemic(22 females, 23 males) and 45 age and sex matched normolipidemic (25 females, 20 males) healhy controls.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group H: Group H: normolipidemic+ periodontally healthy individuals The healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group G: Group G: normolipidemic + gingivitis individuals the healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group CP: Group CP: normolipidemic + generalized chronic periodontitis individuals the healthy controls were randomly selected from among individuals referred to the Periodontology Department for either dental treatment or check-up.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group HH: Group HH: hyperlipidemic + periodontally healthy individuals Hyperlipidemic cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group HG: Group HG: hyperlipidemic + gingivitis individuals Hyperlipidemic cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group HCP: Group HCP: hyperlipidemic + generalized chronic periodontitis individuals Hyperlipidemic cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
Period: Overall Study
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP
Started | 15 | 15 | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group HH: Group HH: hyperlipidemic + periodontally healthy individuals Hyperlipidemic lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group HG: Group HG: hyperlipidemic + gingivitis individuals Hyperlipidemic lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions.
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Group HCP: Group HCP: hyperlipidemic + generalized chronic periodontitis individuals Hyperlipidemic lipid profile and the following cut-off values were used according to the laboratory's recommendation: TC>200mg/dl; TG>200mg/dl; LDL cholesterol >130 mg/dl; HDL <35mg/dl) (29). The diagnosis of the hyperlipidemia had been made at least 3 months before the study, and no distinction was drawn among the hyperlipidemia types. The samples were obtained after a 12-h fasting period from an antecubital vein.
  Periodontal status was assessed by clinical examination and classified according to criteria proposed by the 1999 International World Workshop for a Classification of Periodontal Disease and Conditions
  hyperlipidemia, periodontitis, gingivitis: GCF samples were collected using periopaper strips. Prior to sample collection, each site was gently air-dried, all supragingival plaque was removed, and the area was carefully isolated to prevent samples from being contaminated by saliva
- Total: Total of all reporting groups
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 90
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 38.3 (4.84) | 40.04 (3.93) | 42.17 (3.1) | 45.47 (6.66) | 41 (5.91) | 41.45 (4.81) | 41.40 (4.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 5 | 6 | 7 | 6 | 40
  Male | 7 | 7 | 10 | 9 | 8 | 9 | 50

OUTCOME MEASURES:

1. Primary Outcome: Gingival Crevicular Fluid Level of Malondialdehyde (MDA) as a Marker of Lipid Oxidation.
Description: Malondialdehyde levels in gingival crevicular fluid as measured an oxidative stress marker in lipid. Malondialdehyde (MDA) is the most specific and the most often used molecule in the measurement of biological lipid oxidation
Time Frame: 8-10 am on the day following periodontal status assessment.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
pg/ml | 144.09 (4.15) | 298.52 (18.90) | 802.09 (88.17) | 139.50 (3.40) | 292.98 (4.03) | 899.73 (16.58)

2. Primary Outcome: Protein Carbonyl Level in Gingival Crevicular Fluid as a Marker of Protein Oxidation
Description: Protein carbonylation is another nonenzymatic oxidative post-translational modification and assesed by protein carbonyl tissue content that is often used as a biomarker of oxidative stress.
Time Frame: 8-10 am on the day following periodontal status assessment.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
pg/ml | 0.05 (0.002) | 0.31 (0.004) | 1.91 (0.081) | 0.07 (0.003) | 0.41 (0.019) | 2.89 (0.104)

3. Primary Outcome: Total Antioxidant Capacity Levels in Gingival Crevicular Fluid as a Marker of Antioxidant Status
Description: Contrary to oxidant mediators, TAOC provides an extensive overview of the antioxidant status of the individuals and how well these antioxidants are able to protect host cells during periods of oxidative stress. Due to the potential synergistic effects of different antioxidant molecules, the measurement of TAOC can provide a more accurate and extensive assessment of antioxidant status rather than the separate measurement of individual antioxidant molecules
Time Frame: 8-10 am on the day following periodontal status assessment.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15
pg/ml | 92.21 (1.19) | 78.32 (0.84) | 69.70 (3.37) | 90.32 (0.74) | 70.58 (3.70) | 54.12 (1.06)

ADVERSE EVENTS:
Arm/Group | Group H | Group G | Group CP | Group HH | Group HG | Group HCP
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No